CLINICAL TRIAL: NCT00928642
Title: A Phase II Trial of Gleevec and Gemzar in Patients With Epithelial Ovarian Cancer Who Have Failed at Least Two Prior Therapies
Brief Title: Gleevec and Gemzar in Patients With Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, david mccune, md, Principal Investigator, Madigan Army Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BUS241; MAMC#206126
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer
Keywords: ovarian; cancer; peritoneal; endometrioid; mucinous; serous; clear cell
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Imatinib Mesylate; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Imatinib plus intravenous gemcitabine (Experimental): All research subjects receive oral imatinib 400mg days 1-5 and 8-12 of a 21 day cycle.
  All research subjects received IV gemcitabine 1000mg/m2 days 3 and 10 of a 21-day cycle. .
  All subjects had epithelial ovarian cancer or primary peritoneal carcinomatosis and had failed to respond to prior chemotherapy or progressed after prior chemotherapy.
  Interventions: Drug: imatinib mesylate by mouth; Drug: Gemcitabine Intravenous

INTERVENTIONS:
Drug: imatinib mesylate by mouth — imatinib mesylate - 400mg orally, daily on Days 1-5 and 8-12 of a 21 day cycle.
  Other Names: Gleevec
Drug: Gemcitabine Intravenous — Gemcitabine - 1000 mg/m2 IV on Day 3 and Day 10 of a 21 day cycle
  Other Names: Gemzar

SUMMARY:
This study will evaluate the efficacy and tolerability of the combination of Gleevec and Gemzar in patients with ovarian cancer, who have progressed after receiving at least one prior chemotherapy treatment. Gleevec is an oral chemotherapy drug used is this study and Gemzar is an IV chemotherapy drug used. Participation in the treatment portion of the study will continue as long as the patient's tumors shrink or remain stable and as long as the patient is able to tolerate the study drug. The follow-up portion of the study will last for 5 years.

DETAILED DESCRIPTION:
Each 21 day period will be considered a cycle. Disease status will be assessed with a Cancer Antigen (CA)-125 prior to the start of each new cycle with an assessment of measurable diseased by either CT or MRI every 6 weeks. Treatment will continue until disease progression, unacceptable toxicities, or the patient elects to withdraw from the study. All patients will be followed until disease progression or study withdraw. In addition, following disease progression, patients will be monitored for delayed toxicity and survival for a period of 5 years, unless consent is withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or greater
* Histologically documented diagnosis of ovarian cancer or primary peritoneal cancer. Histological subtypes include: mucinous tumor, serous tumor, endometrioid tumor, and other histologies including clear cell and undifferentiated epithelial tumors.
* At least one measurable site of disease (as defined by Southwestern Oncology Group Solid Tumor Response Criteria) or other response assessment criteria, as appropriate.
* Patients must have relapsed after receiving at least one prior platinum-based chemotherapy.
* Performance status of 0, 1, 2, (ECOG)
* Adequate end organ function: Total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 UNL, creatinine < 1.5 x UNL, ANC > 1.5 x 109/L, platelets > 100 x 109/L.
* Patients will most likely have had their ovaries removed at the time off initial surgery. If any subjects are of childbearing potential at the time of entry, they must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Subjects of reproductive potential must agree to employ and effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of the study drug.
* Written, voluntary informed consent.
* Patients must be eligible for care at a military medical treatment facility.

Exclusion Criteria:

* Patient has received prior treatment with Gemzar.
* Patient has received any other investigational agents within 28 days of the first day of study drug dosing.
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is neither currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Patient with Grade III/IV cardiac problems as defined but the New York Heart Association Criteria.
* Patients who are pregnant or breast-feeding.
* Patient has a severe and/or uncontrolled medical disease (i,e. uncontrolled diabetes, uncontrolled chronic renal disease, or active uncontrolled infection).
* Patient has a known untreated or progressive brain metastasis.
* Patient has known chronic liver diseases (i.e. chronic active hepatitis, and cirrhosis.
* Patient has a known diagnosis of human immunodeficiency virus (HIV infection ).
* Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing..
* Patient previously received radiotherapy to greater than or equal to 25% of the bone marrow.
* Patient had a major surgery within 2 weeks prior to study entry.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David McCune, MD, MPH, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three subjects were enrolled at Brooke Army Medical Center. Five subjects were enrolled at Madigan Army Medical Center.
  Seven of eght subjects are deceased as of 4/4/2013.
Groups:
- Oral Imatinib Plus Gemcitabine: Open label, non-randomized, single treatment group.
Period: Overall Study
Arm/Group | Oral Imatinib Plus Gemcitabine
Started | 8
Completed | 8 (1 subject withdrew after 1st cycle but before disease assessment. 7 of 8 are evaluable for response)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Open label, non-randomized, single treatment group.
Arm/Group | Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: The Cystostatic, Anti-tumor Activity of the Combination of Gleevec and Gemzar Via Progression-free Survival for at Least Six Months in Patients With Recurrent or Persistent Epithelial Ovarian or Primary Peritoneal Carcinoma.
Description: Progression free survival at six months was assessed for all research subjects. Progression defined by SWOG criteria: Invest New Drugs. 1992 Nov;10(4):239-53. Progression is defined as > 50% increase in the sume of measured cross sectional area of areasa of measurable disease, measured from the lowest measured amount of disease. Progression is also defined as new areas of measurabe disease.
Time Frame: Time to progression was measured from enrollment in study until documented disease progression over a period not greater than 2 years.
Population: of 8 enrolled subjects, 7 were eligible for analysis of progression-free survival at 8 months. One subject declined to continue treatment
Measure: Number; unit: participants
Groups:
- Oral Imatinib Plus Gemcitabine: Open label, non-randomized, single treatment group.
  All subjects has measurable or evaluabel epithelial ovarian cancer or preitoneal carcinomatosis. all subjects were treated with oral imatinib and IV gemcitabine.
Arm/Group | Oral Imatinib Plus Gemcitabine
Number analyzed (Participants) | 7
participants | 0

2. Primary Outcome: To Determine the Safety and Tolerability Via Frequency and Severity of Adverse Effect of Combination Gleevec and Gemzar in This Cohort of Patients as Assessed Byt Common Toxicity Criteria
Description: Toxicity was assess prior to each cycle of therapy (every 3 weeks) and graded based on NCI common toxicity criteria
Time Frame: Until disease progression or unacceptable toxicity
Measure: Number; unit: participants
Groups:
- Oral Imatinib Puls IV Gemcitabine: Open label, non-randomized, single treatment group.
Arm/Group | Oral Imatinib Puls IV Gemcitabine
Number analyzed (Participants) | 8
participants
  Grade 3 toxicity | 3
  Grade 4 toxicity | 1
  Red Blood Cell Transfusion | 1

3. Secondary Outcome: Tumor Response Rates Using Modified SWOG Criteria to the Combination of Gleevec and Gemzar in Patients With Relapsed Ovarian Cancer Who Have Failed at Least One Prior Chemotherapy Treatment.
Description: Best response to thearpy was assessed using modified SWOG criteria (same as for outcome masure #1). Subjects were assess as "complete response", "partial response", "stable disease", and "progressive disease" after 2 cycles (6 weeks) of beginning treatment and every 6 weeks afterward until progression of disease, unacceptable toxicity, or subject withdrawl from study.
  the measurement reported is the number of patients who met the criteria for partial response.
Time Frame: Subjects treated until progression of disease or unacceptable toxicity. no maximum dose was specified
Population: All subjects who underwent treatment and participated in the study were analysed
Measure: Number; unit: participants
Groups:
- Oral Imatinib Plus IV Gemcitabine: Open label, non-randomized, single treatment group. all subjects had epithelial ovarian cancer or primary peritoneal carcinomatosis that progressed after prior treatment.
Arm/Group | Oral Imatinib Plus IV Gemcitabine
Number analyzed (Participants) | 7
participants | 0

4. Secondary Outcome: To Determine the Distribution of the Overall Survival
Description: All subjects were followed after treatment was complete to assess overall survival.
Time Frame: Until death
Measure: Median (Full Range); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 8
months | 9 [2 to 41]

5. Secondary Outcome: To Estimate the Clinical Response Rate(Partial and Complete Response as Defined Under the SWOG Criterial)
Description: Using SWOG criteria for response of measurable disease, subject best response was assessed. First assessment was 6 weeks after starting treatment. Subjequent evaluations were every 6 weeks in patients who remained on study.
  Repsonse rate was the sum of Complete Repsonse and Partial Response.
Time Frame: until disease progression or unacceptable toxicity
Population: All subjects were assessed after 6 weeks of treatment and reassessed at 6 week intervals
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 7
participants | 0

6. Secondary Outcome: To Assess the Effects of Prognostic Variables; Initial Performance Status; Platinum Sensitivity, and Mucinous (or Clear Cell)Histology on Progression-free Survival Overall.
Description: The study was stopped after 8 subjects. It was not possible to perform meaningful analysis on prognostic variables. this outcome measure was not done.
Time Frame: Until disease progression
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from initiation of treatment to 30 days off treatment.
Description: Adverse events were scored based on NCI common toxicity criteria. All serious adverse events and all non-serious adverse events were reported.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Cellulitis of the leg developed, resolved with appropriate antibiotics and no sequelae
Pyelonephritis (Renal and urinary disorders) | 1 (1) — One subject pyelonephritis that was possibly study related and responded to treatment.
Allergic Reaction (Immune system disorders) | 1 (1) — One subject develoed tongue swelling after cycle #1. Treatment was discontinued and no other episodes were observed
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 4 neutropenia - treated with dose reduction

LIMITATIONS AND CAVEATS:
This study was terminated due to a combination of poor accrual and lack of evidence of benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No